CLINICAL TRIAL: NCT00995566
Title: Thelin (Sitaxentan Sodium) Patient Safety Registry A Non-Interventional, Patient Registry For The Collection Of Pre-Defined Safety Data In Patients Prescribed Thelin
Brief Title: A Non-Interventional, Patient Registry For The Collection Of Pre-Defined Safety Data In Patients Prescribed Thelin
Acronym: PROSE
Status: Terminated | Type: Observational
Why Stopped: The trial was prematurely terminated on Dec 9, 2010, due to safety concerns, specifically new emerging evidence of hepatic injury."
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Other Study IDs: B1321045
Record Dates: First submitted 2009-09-17; First posted 2009-10-15 (Estimated); Results first posted 2012-02-01 (Estimated); Last update posted 2012-02-07 (Estimated); Status verified 2011-05

CONDITIONS: Pulmonary Arterial Hypertension
MeSH Terms: conditions — Pulmonary Arterial Hypertension

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Thelin Registry Patients
  Interventions: Drug: Sitaxentan sodium

INTERVENTIONS:
Drug: Sitaxentan sodium — Please note that this is a non-interventional study and no drug is actually given as an intervention. Instead, patients prescribed THELIN are being followed under real world circumstances. However at the request of the QA group at CT.gov, we were instructed to add sitaxentan sodium as the intervention type, regardless of the fact that this is a non-interventional study.

SUMMARY:
The Thelin Patient Safety Registry is a post-marketing program in the European Union (EU) that is designed to supplement the reporting of spontaneous adverse events (AE) and better characterize known and potential safety signals for Thelin. The registry is a secure, restricted access, electronic system which collects anonymous, pre-defined, patient-level data on demographic variables, safety monitoring measurements (i.e. liver function tests, haemoglobin and international normalized ratio (INR) measurements), concomitant medications, information on AEs and Thelin drug discontinuation. Regular review of the data is conducted to assess the frequency of identified safety risks and to monitor for the emergence of new safety signals at monthly pharmacovigilance meetings, quarterly signal detection meetings, and for each Periodic Safety Update Report (PSUR).

DETAILED DESCRIPTION:
Non-probability sample

ELIGIBILITY:
Inclusion Criteria:

* Evidence of a personally signed and dated informed consent document by the patient indicating that he/she (or a legally acceptable representative) has been informed of all pertinent aspects of the study is a requirement for inclusion.
* Additional inclusion criteria reflect the approved label for Thelin as outlined in the SmPC.

Exclusion Criteria:

* There are no specific exclusion criteria for enrollment in the Thelin Patient Safety Registry, with the exception of those reflected in the approved label for Thelin as outlined in the SmPC.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: * All patients enrolled must meet the usual prescribing criteria for Thelin as per the Summary of Product Characteristics (SmPC) and are enrolled in the registry at the clinician's discretion.
  * All prescribers are offered the opportunity to participate in the registry, assuming they have received appropriate educational materials
Sampling Method: Non-Probability Sample
Enrollment: 54 (Actual)
Dates: Start 2010-04; Primary Completion 2011-02 (Actual); Study Completion 2011-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (4):
- Belgium (2):
  - Pfizer Investigational Site, Brussels
  - Pfizer Investigational Site, Leuven
- Pfizer Investigational Site, Nice, France
- Pfizer Investigational Site, Hanover, Germany

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=B1321045&StudyName=A%20Non-Interventional%2C%20Patient%20Registry%20For%20The%20Collection%20Of%20Pre-Defined%20Safety%20Data%20In%20Patients%20Prescribed%20Thelin%20

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The Sitaxentan Sodium program was discontinued December 10, 2010.
Groups:
- Thelin Registry Patients: The use and dosage recommendations for Thelin (sitaxentan sodium) was in accordance with the local summary of Product Characteristics.
Period: Overall Study
Arm/Group | Thelin Registry Patients
Started | 54
Completed | 0
Not Completed | 54
Not completed — Adverse Event | 2
Not completed — Early study termination | 52

BASELINE CHARACTERISTICS:
Arm/Group | Thelin Registry Patients
Number analyzed (Participants) | 54
Age Continuous [Mean (Standard Deviation); unit: years] | 60.5 (18.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 41
  Male | 13

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Elevated Liver Function Post-baseline
Description: Elevated liver function: greater than 3 times the upper limit of normal (>3 x ULN) alanine aminotransferase (ALT) and aspartase aminotransferase (AST) levels. Laboratory data were analyzed by several local laboratories. There were subtle differences in the reference ranges used for analyses.
Time Frame: Monthly up to 1 year
Population: Full Analysis Set (FAS): participants enrolled in Patient Registry of Sitaxentan in Europe (PROSE). Number of participants analyzed (N): participants with evaluable data.
Measure: Number; unit: percentage of participants
Arm/Group | Thelin Registry Patients
Number analyzed (Participants) | 45
percentage of participants
  ALT >3 xULN | 2.2
  AST >3 xULN | 2.2

2. Primary Outcome: Percentage of Participants With a Decrease in Hemoglobin Post-baseline
Description: Laboratory data were analyzed by several local laboratories. There were subtle differences in the reference ranges used for analyses.
Time Frame: Monthly up to 1 year
Population: Data not summarized due to the small number of participants in database.
Measure: Number; unit: percentage of participants
Arm/Group | Thelin Registry Patients
Number analyzed (Participants) | 0

3. Primary Outcome: Percentage of Participants With Increases in Total, Conjugated and Non-conjugated Bilirubin Post-baseline
Description: Total and conjugated bilirubin levels measured from blood, but indirect bilirubin calculated. Indirect bilirubin=Total bilirubin - Conjugated bilirubin. Laboratory data were analyzed by several local laboratories. There were subtle differences in the reference ranges used for analyses.
Time Frame: Monthly up to 1 year
Population: Data not summarized due to the small number of participants in database.
Measure: Number; unit: percentage of participants
Arm/Group | Thelin Registry Patients
Number analyzed (Participants) | 0

4. Primary Outcome: Duration of Exposure to Thelin
Description: Time between the first and last dose of Thelin. For participants who continued Thelin from TOPS (another study), the initial TOPS' Thelin start date was used.
Time Frame: 1 Year
Population: FAS
Measure: Mean (Standard Deviation); unit: months
Arm/Group | Thelin Registry Patients
Number analyzed (Participants) | 54
months | 21.5 (15.3)

5. Primary Outcome: Adverse Events (AEs) by Seriousness and Relationship to Treatment
Description: Counts of participants who had AEs or treatment-emergent adverse events (TEAEs), defined as newly occurring or worsening after first dose. Serious adverse events (SAEs) were reported from the time of informed consent. Relatedness to Thelin was assessed by the investigator (Yes/No). Participants with multiple occurrences of an AE within a category were counted once within the category.
Time Frame: Baseline up to year 1
Population: FAS
Measure: Number; unit: participants
Arm/Group | Thelin Registry Patients
Number analyzed (Participants) | 54
participants
  Any TEAE | 11
  TEAE related to Thelin | 1
  SAE | 6
  SAE related to Thelin | 1

6. Primary Outcome: Clinical Status Since Last Visit
Description: Clinical status determined by status of pulmonary arterial hypertension (PAH) since last visit, reported as PAH remained stable, improved or deteriorated.
Time Frame: Monthly up to 1 year
Population: Data not summarized due to the small number of participants in database.
Measure: Number; unit: participants
Arm/Group | Thelin Registry Patients
Number analyzed (Participants) | 0

7. Primary Outcome: Concomitant Medications
Description: Number of participants with concomitant medication usage reported by drug categories.
Time Frame: Baseline, monthly up to 1 year
Population: Data not summarized due to the small number of participants in database.
Measure: Number; unit: participants
Arm/Group | Thelin Registry Patients
Number analyzed (Participants) | 0

8. Primary Outcome: Bleeding AEs by Seriousness, Relationship to Treatment, Endothelin-A Receptor Antagonist (ERA) Usage, and International Normalized Ratio (INR) Results
Description: Counts of participants who had bleeding events or treatment-emergent bleeding events, defined as newly occurring or worsening after first dose. Serious bleeding events reported from time of informed consent. Relatedness to Thelin assessed by investigator (Yes/No). ERA usage: was participant taking Vitamin K antagonist? (Yes/No). INR: participant's prothrombin time (PT) ratio. Participants with multiple occurrences of an AE within a category were counted once within the category.
Time Frame: Baseline up to year 1
Population: FAS
Measure: Number; unit: participants
Arm/Group | Thelin Registry Patients
Number analyzed (Participants) | 54
participants
  Any bleeding event | 1
  Bleeding event related to Thelin | 0
  Serious bleeding event | 0
  Serious bleeding event related to Thelin | 0
  Bleeding event with ERA usage | 0
  Bleeding event with INR results | 0

9. Primary Outcome: Percentage of Participants Who Experienced Pulmonary Edema With the Presence of Veno-occlusive Disease
Description: The criteria used to determine whether participants had both pulmonary edema and veno-occlusive disease was at the discretion of the Investigator.
Time Frame: Baseline up to year 1
Population: FAS
Measure: Number; unit: percentage of participants
Arm/Group | Thelin Registry Patients
Number analyzed (Participants) | 54
percentage of participants | 0

ADVERSE EVENTS:
Description: The same event may appear as both an AE and a SAE. However, what is presented are distinct events. An event may be categorized as serious in 1 participant and as nonserious in another participant, or 1 participant may have experienced both a serious and nonserious event during the study.
Arm/Group | Thelin Registry Patients
Serious Adverse Events (participants affected / at risk) | 6/54
Other Adverse Events (participants affected / at risk) | 6/54
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Thelin Registry Patients (N=54)
Cardiac failure (Cardiac disorders) | 3
Hyperparathyroidism primary (Endocrine disorders) | 1
Oedema (General disorders) | 1
Hepatitis toxic (Hepatobiliary disorders) | 1
Injection site infection (Infections and infestations) | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1
Paraesthesia (Nervous system disorders) | 1
Agitation (Psychiatric disorders) | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary arterial hypertension (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Thelin Registry Patients (N=54)
Atrial tachycardia (Cardiac disorders) | 1
Anal haemorrhage (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 1
Chest pain (General disorders) | 1
Arthritis (Musculoskeletal and connective tissue disorders) | 1
Headache (Nervous system disorders) | 1
Hypotension (Vascular disorders) | 1

LIMITATIONS AND CAVEATS:
The protocol did not identify the priority of endpoints. Therefore, all endpoints arbitrarily assigned as primary.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.